CLINICAL TRIAL: NCT06643325
Title: Gastric Point-of-care Sonography with Focus on Gastric Emptying Time in Patients with Traumatic Injuries. a Prospective Observational Study
Brief Title: Gastric Emptying Time in Traumatic Injuries
Status: Recruiting | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Other Study IDs: POCUS 2
Record Dates: First submitted 2023-04-03; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia; Gastric Ultrasound; Sonography; Point of Care Ultrasound (POCUS); Regurgitation; Pulmonary Aspiration During Anesthetic Induction; Trauma Patients
Keywords: point of care ultrasound; gastric ultrasound; trauma patients; aspiration; anesthesia
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Gastric ultrasound — Serial, gastric sonography

SUMMARY:
The investigators plan to do serial sonographic examinations of the gastric antrum (quantity, quality) to estimate the gastric emptying time and dependant factors after traumatic injurys.

DETAILED DESCRIPTION:
The investigators plan to do serial sonographic examinations of the gastric antrum (quantity, quality) in patients suffering from a relevant traumatic injury. Patients which are admitted to the emergency department with a corresponding history are considered for inclusion. Patient with life-threatening injuries are excluded. After inclusion, the investigators plan to carry out gastric ultrasound (POCUS) all 2 hours until the operative treatment (maximal 5 examinations). To identify factors which may be correlated with delayed gastric emptying several demographic and patient related factors are collected.

ELIGIBILITY:
Inclusion Criteria:

* relevant traumatic injury

Exclusion Criteria:

* life-threatening traumatic injury (immediate treatment is necessary)
* Underage
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the emergency department with a relevant traumatic injury
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Sonographic quality/quantity of the gastric antrum | 2 hour
  Quality of the gastric content (empty, fluid, solid or mixed fluid/solid) and quantity of the gastric content in ml, measured in 2 hour time intervals

SECONDARY OUTCOMES:
Pain-scale | 2 hour
  Evaluate pain using the VAS Scale 0-10 (Visual Analog Scale)
Analgetics | 2 hour
  Evaluate need of analgetics
Stress, activation of sympathic nerve system | 2 hour
  Evaluate stress on a VAS 0-10 (Visual Analog Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Winterthur, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided